CLINICAL TRIAL: NCT06583850
Title: Evaluation of Pain, Cervical Mobility, Sleep Quality and Functional Status in Individuals with Chronic Neck Pain
Brief Title: Chronic Neck Pain: Mobility, Sleep, Function
Acronym: observational
Status: Completed | Type: Observational
Sponsor: Gamze Demircioğlu (Other)
Responsible Party: Sponsor-Investigator, Gamze Demircioğlu, Principal Investigator, Atlas University
Organization: Atlas University (Other)
Other Study IDs: neckpain
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Pain; Neck
Keywords: pain; neck; range of motion; sleep quality; functional status
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- chronic neck pain: chronic neck pain (CNP) (persists longer than 3 months.
  Interventions: Other: The Neck Disability Index; Other: Visual analog scale (VAS); Other: Pittsburgh Sleep Quality Index; Other: Cervical Range of Motion Assessment
- control: healthy controls
  Interventions: Other: The Neck Disability Index; Other: Visual analog scale (VAS); Other: Pittsburgh Sleep Quality Index; Other: Cervical Range of Motion Assessment

INTERVENTIONS:
Other: The Neck Disability Index — The Neck Disability Index (NDI) is the most widely used self-report tool to assess neck pain status, and provides information not only about pain experiences but also about a person's functional status. The NDI consists of 10 questions related to pain, functional activities, self-care, and quality of life that are measured on a 6-point scale (0, no disability; 5, full disability). The numeric score for each item is summed for a score ranging from 0 to 50; 0-4 points are defined as no disability, 5-14 points as mild disability, 15-24 points as moderate disability, 25-34 points as severe disability and above 35 points as complete disability.
Other: Visual analog scale (VAS) — A 10 cm VAS numbered from 0 to 10 was used for the assessment. 0 indicates no pain and 10 indicates unbearable pain. Participants were asked to mark a point between 0-10 according to their pain status
Other: Pittsburgh Sleep Quality Index — Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-report questionnaire
Other: Cervical Range of Motion Assessment — Active Cervical Range Of Motion was measured with a universal goniometer in all three planes of motion in the cervical region: lateral flexion (frontal plane), axial rotation to both right and left sides (horizontal plane), and flexion-extension (sagittal plane).

SUMMARY:
The goal of this observational study is to compare pain, cervical mobility, sleep quality, and functional status between individuals with chronic neck pain (CNP) and healthy individuals. The study focuses on understanding the complex relationships between these factors in individuals with CNP, with the aim of providing insights that could contribute to more effective rehabilitation strategies.

The main questions it aims to answer are:

* How pain, cervical mobility, sleep quality, and functional status differs between individuals with and without chronic neck pain?
* What is the relationship between functional status and cervical mobility and sleep quality in individuals with chronic neck pain?

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years.
* Chronic neck pain (CNP) persisting for longer than 3 months (for the CNP group).
* Volunteering participation in the study.
* Healthy controls, including relatives of CNP participants.

Exclusion Criteria:

* History of neck trauma or other cervical spine conditions (e.g., radiculopathy).
* Prior surgical interventions involving the head, face, cervical spine, upper or lower extremities, or cervical disc herniation.
* Degenerative spinal conditions.
* Use of analgesics, anti-inflammatory medications, or muscle relaxants within the previous week.
* Presence of rheumatological or cardiovascular diseases, chronic neurological or psychiatric disorders, substance abuse, anemia, or diabetes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chronic neck pain and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
The Neck Disability Index | Baseline
  The Neck Disability Index (NDI) is the most widely used self-report tool to assess neck pain status, and provides information not only about pain experiences but also about a person functional status. The NDI consists of 10 questions related to pain, functional activities, self-care, and quality of life that are measured on a 6-point scale (0, no disability; 5, full disability). The numeric score for each item is summed for a score ranging from 0 to 50; 0-4 points are defined as no disability, 5-14 points as mild disability, 15-24 points as moderate disability, 25-34 points as severe disability and above 35 points as complete disability.
Pittsburgh Sleep Quality | Baseline
  Five questions on the scale are answered by the participant's partner or roommate and are used solely for clinical information..The PSQI has seven components: subjective sleep quality, sleep latency, total sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The total score is calculated by summing the scores of the seven components, ranging from 0 to 21 points.
Visual analog scale | Baseline
  A 10 cm VAS numbered from 0 to 10 was used for the assessment. 0 indicates no pain and 10 indicates unbearable pain.
Range of motion | Baseline
  Active Cervical Range of Motion Assessment was measured with a universal goniometer in all three planes of motion in the cervical region: lateral flexion (frontal plane), axial rotation to both right and left sides (horizontal plane), and flexion-extension (sagittal plane). The same physiotherapist performed all goniometric measurements to eliminate any differences between the measurements that the measurer could cause. The American Association of Orthopaedic Surgeons (AAOS) values were taken as a reference for NEH in the cervical region. Care was taken to ensure that the participant wore comfortable clothes during the measurements. Before starting the measurement, the desired movement was shown to the participant by the physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas Univercity, Istanbul, Hamidiye, Turkey (Türkiye)